CLINICAL TRIAL: NCT00048594
Title: A Double-Blind, Placebo-Controlled, Multicenter Study of the Long-Term Efficacy of MK0869 in the Maintenance of Antidepressant Effect in Patients With Major Depressive Disorder
Brief Title: Long Term Treatment of Patients With Major Depressive Disorder With MK0869 (0869-065)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-065; Formally-35MRB2; MK0869-065; 2006_405
Record Dates: First submitted 2002-11-04; First posted 2002-11-05 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: aprepitant
  Other Names: MK0869
Drug: Comparator: placebo (unspecified)

SUMMARY:
A clinical study to determine the efficacy and safety of an investigational medication (MK0869) in the treatment of depression.

DETAILED DESCRIPTION:
The duration of treatment is 20 months.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2002-01-03 (Actual); Primary Completion 2003-12-18 (Actual); Study Completion 2003-12-22 (Actual)

PRIMARY OUTCOMES:
Total HAMD-17 score </= 10 after 10 weeks of treatment, time to relapse of depression over 6-10 months | after 10 weeks of treatment and over 6-10 months

SECONDARY OUTCOMES:
CGI-S score change from Week 10 at Month 6; HAMD-17 total score change from Week 10 at Month 6; an HAMA total score change from week 10 at Month 6. | Week 10 at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/policies-perspectives.html